CLINICAL TRIAL: NCT04450940
Title: Examining the Impact of PACV Administration on Vaccine Hesitancy: a Randomized Control Trial, Houston, TX
Brief Title: Impact of PACV Administration on Vaccine Hesitancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Julie Boom, Medical Director, Immunization Project; Associate Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: H33255
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Evaluating Impact of PACV on Vaccine Hesitancy Among Parents of Newborns
Keywords: Parental Attitudes about Childhood Vaccines; vaccine hesitancy
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: Participants were randomized to receive 1 of 2 surveys at enrollment - either the PACV (a survey that identifies vaccine hesitant parents) or a placebo survey on general childhood health topics. 6 months following enrollment, all participants received the PACV, regardless of baseline randomization group.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Clinic staff, study authors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACV (Experimental): The PACV arm received the PACV survey at baseline in order to assess the impact of administration on vaccine hesitancy. All participants received the PACV at 6-month follow up.
  Interventions: Behavioral: PACV survey
- Placebo (Sham Comparator): The placebo arm received a placebo survey on general childhood health topics at baseline. All participants received the PACV at 6-month follow up.
  Interventions: Behavioral: Placebo survey

INTERVENTIONS:
Behavioral: PACV survey
  Arms: PACV
Behavioral: Placebo survey
  Arms: Placebo

SUMMARY:
Our objective is to assess the impact of administering the PACV to parents of newborns. We also sought to assess the prevalence of vaccine hesitancy among parents of newborns in Houston, TX and to characterize the demographics of vaccine-hesitant parents.

DETAILED DESCRIPTION:
Despite overwhelming scientific evidence demonstrating the safety and effectiveness of vaccines, parental immunization concerns continue to increase. Compared to parents who refuse all vaccines, vaccine-hesitant parents (VHP), defined as parents who are ambivalent towards vaccines, are of particular interest because they tend to be more amenable to vaccination. VHPs tend to be part of a larger group of parents with moderate vaccine concerns who seek additional information from their healthcare provider before deciding whether or not to immunize. These parents will sometimes immunize after education and reassurance from their provider. Alternatively, they may choose to delay or refuse certain vaccines. It is important to identify VHPs early in the medical relationship to provide effective communication and appropriate education regarding vaccine concerns in order to ensure maximum immunization coverage for the children of these parents.

The Parent Attitudes about Childhood Vaccines (PACV) survey was previously developed to identify VHPs. In a follow up study, the survey was validated and found to be a reliable instrument in identifying VHPs. The PACV survey differs from other survey instruments in that it seeks to specifically identify VHPs. Moreover, the survey was found to be a reliable predictor of immunization status with higher total PACV scores associated with under-immunization.5 It is unknown if administering the PACV survey can have a negative impact on parental immunization beliefs or if the PACV survey can elicit vaccine concerns that otherwise would not have been present at that point in time.

Study enrollment will occur among parents/guardians of children who are scheduled at a Texas Children's Pediatric practice for an 2-week well child visit. Parents/guardians of children will receive an enrollment packet containing a self-screening form, cover letter, and survey from the practice staff at their appointment check-in. Parents will be randomized to receive 1 of 2 surveys - either the PACV or a placebo survey about general childhood health topics. Upon receipt of the enrollment packet, the parent/guardian will be asked to complete a self-screening form to determine if they meet eligibility criteria. If the parent/guardian does not meet eligibility criteria the self-screening form will direct them to return the enrollment packet unopened to the front desk staff. Parents/guardians of children meeting eligibility criteria will be directed to open the enrollment packet and complete the survey. The PACV survey will then be administered to all subjects six months following the initial survey administration.

Prevalence of vaccine hesitancy will be calculated for each group (initial PACV or placebo survey) separately and then for both groups combined. PACV scores calculated from the second administration at 6 months will be compared across groups to evaluate if administration of the PACV increases vaccine hesitancy.

Inclusion criteria:

1. Person must self-identify as English-speaking.
2. Parent of a child less than 3 months of age.
3. Parent must be 18 years of age or older.
4. Parent of a child seeking routine, well-child care at a selected TCP practice site.

Exclusion criteria:

1. Person does not self-identify as English-speaking.
2. Parent of child greater than 3 months of age.
3. Parent is less than 18 years of age.
4. Parent of child not seeking routine, well-child care at a selected TCP practice site.

ELIGIBILITY:
Inclusion Criteria:

1. Person must self-identify as English-speaking.
2. Parent of a child less than 3 months of age.
3. Parent must be 18 years of age or older.
4. Parent of a child seeking routine, well-child care at a selected TCP practice site.

Exclusion Criteria:

1. Person does not self-identify as English-speaking.
2. Parent of child greater than 3 months of age.
3. Parent is less than 18 years of age.
4. Parent of child not seeking routine, well-child care at a selected TCP practice site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1705 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Impact of PACV administration on vaccine hesitancy | 6 months
  We assessed the change in the proportion of vaccine-hesitant parents between baseline and 6-month follow up

SECONDARY OUTCOMES:
Prevalence of vaccine hesitancy | 6 months
  We assessed the proportion of vaccine-hesitant parents
Summarize characteristics of vaccine-hesitant parents | 6 months
  We sought to summarize the demographic characteristics of vaccine-hesitant parents and examine associations between vaccine hesitancy and participant characteristics

IPD SHARING:
Plan to Share IPD: No